CLINICAL TRIAL: NCT03878355
Title: Long-term Outcomes of Radical Endoscopic Sinus Surgery Plus Draf 3 Procedure in Eosinophilic Chronic Rhinosinusitis With Nasal Polyps and Asthma: A 9-year Prospective Study
Brief Title: A Study of Different Endoscopic Surgery Procedures in Eosinophilic Chronic Rhinosinusitis With Nasal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-ES
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Surgery
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned 1:1:1 to receive FESS, RESS and RESS plus Draf 3 surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- radical endoscopic sinus surgery plus Draf 3 surgery (Experimental)
  Interventions: Procedure: radical endoscopic sinus surgery (RESS) plus Draf 3 surgery.
- radical endoscopic sinus surgery (Experimental)
  Interventions: Procedure: radical endoscopic sinus surgery (RESS)
- functional endoscopic sinus surgery (Experimental)
  Interventions: Procedure: functional endoscopic sinus surgery (FESS)

INTERVENTIONS:
Procedure: radical endoscopic sinus surgery (RESS) plus Draf 3 surgery. — The procedure of RESS was completed as described in "full-house FESS (FHF)" approach, involving complete removal of all nasal polyps along with a full maxillary antrostomy, total ethmoidectomy, wide sphenoidotomy, and a Draf 2A frontal sinusotomy. Moreover the bilateral inferior two-thirds of MTs were meanwhile resected. The technique for the Draf 3 frontal drillout procedure was described in detail in previous publications with resection of the superior nasal septum, central frontal sinus floor, and frontal beak region, resulting in a widely patent, oval-shaped, common frontal sinus neo-ostium
  Arms: radical endoscopic sinus surgery plus Draf 3 surgery
Procedure: radical endoscopic sinus surgery (RESS) — The procedure of RESS was completed as described in "full-house FESS (FHF)" approach, involving complete removal of all nasal polyps along with a full maxillary antrostomy, total ethmoidectomy, wide sphenoidotomy, and a Draf 2A frontal sinusotomy. Moreover the bilateral inferior two-thirds of MTs were meanwhile resected
  Arms: radical endoscopic sinus surgery
Procedure: functional endoscopic sinus surgery (FESS) — FESS was performed by Messerklinger technique with middle turbinate preservation
  Arms: functional endoscopic sinus surgery

SUMMARY:
CRS remains a common challenging clinical entity due to variable phenotypes with different underlying mechanisms that lead to persistence or recurrence polyps. The eosinophils dominant inflammation was considered as a major pathological hallmark and challenges of CRS with nasal polyps (CRSwNP). Differentiate surgical approaches towards eosinophilic CRSwNP (eCRSwNP) should be addressed on the basis of the inflammatory endotypes. eCRSwNP has been recognized as the most easily relapsed type of CRS, and the combination of asthma increases the difficulty of treatment. Till now there is no recognized surgical strategy for eCRSwNP with asthma.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of CRSwNP was based on the standard criteria issued in the European Position Paper on Rhinosinusitis and Nasal Polyps guidelines.
* Participants had at least 1 previous sinus surgery underwent FESS (middle turbinate (MT) preserved), good gasification of frontal sinus and with concomitant asthma.
* The diagnosis of asthma was confirmed by a chest physician according to Global Initiative for Asthma (GINA) guidelines.
* Polyp biopsy was undertaken 1 week before surgery and the eCRSwNP was confirmed by the number of eosinophils exceeded 10% of total infiltrating inflammatory cells in the polyp tissue through the evaluation by using hematoxylin and eosin (H&E) staining.

Exclusion Criteria:

* Patients were excluded if they had unilateral disease, allergic fungal rhinosinusitis, antrochoanal polyps, or cysts.

Ages: 24 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
recurrence | 1 year after surgery
  Recurrence was defined if the patient had symptoms of chronic rhinosinusitis after surgery, and nasal endoscopy found nasal polyps recurrence, obvious edema of mucosa, or purulent secretion, and above of symptoms or physical signs existed, which can't be alleviated by maximum medicine treatment at least 1 month
recurrence | 3 years after surgery
  Recurrence was defined if the patient had symptoms of chronic rhinosinusitis after surgery, and nasal endoscopy found nasal polyps recurrence, obvious edema of mucosa, or purulent secretion, and above of symptoms or physical signs existed, which can't be alleviated by maximum medicine treatment at least 1 month
recurrence | 5 years after surgery
  Recurrence was defined if the patient had symptoms of chronic rhinosinusitis after surgery, and nasal endoscopy found nasal polyps recurrence, obvious edema of mucosa, or purulent secretion, and above of symptoms or physical signs existed, which can't be alleviated by maximum medicine treatment at least 1 month

SECONDARY OUTCOMES:
Visual analogue scale of 4 major clinical symptoms | at baseline, and 1 year, 3years, 5 years after surgery
  Subjective symptoms were scored on a visual analogue scale of 0 to 10 as previously described, with 0 being no complaints whatsoever and 10 being the worst imaginable. Four major symptoms include nasal congestion, rhinorrhea, loss of smell, and headache and/or facial pain.
Sinus-specific quality of life (QoL) | at baseline, and 1 year, 3years, 5 years after surgery
  Sinus-specific quality of life (QoL) was assessed using the 22-item Sinonasal Outcome Test (SNOT-22)
Postoperatively endoscopic results | at baseline, and 1 year, 3years, 5 years after surgery
  Postoperatively endoscopic results were scored according to the Lund-Kennedy system, with the assessment of edema, nasal discharge, scarring, and crusting